CLINICAL TRIAL: NCT04390659
Title: Myomectomy During Cesarean Section,Is This Aright Decision
Brief Title: Myomectomy During Cesarean Section Is This Aright Decision
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, clinical professor, Benha University
Other Study IDs: khalid7
Record Dates: First submitted 2020-04-29; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Obstetric Labor, Premature
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Uterine Myomectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: myomectomy — The myomectomy was done by conventional technique but timing of myomectomy either before or after delivery of the baby varied between different cases .Infusion of oxytocin during the operation and for 24 h later.

SUMMARY:
myomectomy was done during cesarean section

DETAILED DESCRIPTION:
The myomectomy was done by conventional technique but timing of myomectomy either before or after delivery of the baby varied between different cases .Infusion of oxytocin during the operation and for 24 h later.

ELIGIBILITY:
Inclusion Criteria:

* women with diagnosed uterine myoma prior to pregnancy
* needed cesarean sections for various indications.
* Women with diagnosed uterine myoma during pregnancy and needed cesarean sections for various indications.
* Women with myoma diagnosed incidentally during labour.

Exclusion Criteria:

* Refusal of the women at any time before and during the operations.
* Cervical myoma.
* Atonic uterus after delivery of the baby.
* Women with bleeding disorders due to medical or obstetric causes.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: c s with uterine myoma
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
difficulty of cesarean myomectomy | during the procedure/surgery"
  according to the site and type of myoma

SECONDARY OUTCOMES:
4concentrations of hemoglobin | during the procedure
  intra operative bleeding

CONTACTS AND LOCATIONS:
Overall Officials: khalid salama, Principal Investigator — Benha University

IPD SHARING:
Plan to Share IPD: No
master sheet

REFERENCES:
- [Result] Ledee-Bataille N, Lapree-Delage G, Taupin JL, Dubanchet S, Frydman R, Chaouat G. Concentration of leukaemia inhibitory factor (LIF) in uterine flushing fluid is highly predictive of embryo implantation. Hum Reprod. 2002 Jan;17(1):213-8. doi: 10.1093/humrep/17.1.213. PMID 11756390